

| Document Title: | Statistical Analysis Plan BIO Master.BIOMONITOR III |
|---|---|
| Document Version and Date: | Version 3-0, 15-June-2022 |
| ClinicalTrials.gov Identifier: | NCT04025710 |

Sponsor:

Rev. B

| BIOTRONIK SE & Co. KG |
|------------------------------------|
| BIO MASTER.BIOMONITOR III / BA 109 |

| • | |
|---|---|
| Study name / EAC code: | BIO MASTER.BIOMONITOR III / BA 109 |
| Version and date of the Statistical Analysis Plan: | Version 3.0 from 15 JUN 2022 |
| Version and date of the underlying<br>Clinical Investigation Plan: | Version 1.0 from 12 JUL 2019 |

| Print Name & Title | Signature | Date of Signature (DD MMM YYYY) |
|--------------------|-----------|---------------------------------|
| Project Manager | | |
| Scientists | | 21 JUN 2022 |
| Biostatistician | | 21 JUN 2022 |

by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality:

This document and/or its contents are only for internal use.

# **Table of Content**

| Table of Content | 2 |
|-------------------------------------------------------------|----|
| 1. Introduction | 4 |
| 1.1. Aim | 4 |
| 1.2. General information | 4 |
| 2. Objectives | 6 |
| 3. Investigational Device | 6 |
| 4. Study Design & Time Course | 6 |
| 5. General Statistical Procedures | 8 |
| 5.1. Descriptive analyses | 8 |
| Nominal – dichotomous data | 8 |
| Nominal data – more than two categories | 8 |
| Scale / metric data | 9 |
| Ordinal data | 9 |
| 5.2. Inferential analyses | 10 |
| 5.3. Significance level | 10 |
| 5.4. Missing Data | 10 |
| 5.5. Exclusion of data from confirmatory data analysis | 10 |
| 5.6. Subgroups | 11 |
| 5.7. Interim analyses | 11 |
| 5.8. Software | 12 |
| 6. Specific Study Dates | 13 |
| 6.1. Enrollment date | 13 |
| 6.2. Insertion date | 13 |
| 6.3. Termination date | 13 |
| 7. Analysis Sets | 14 |
| 7.1. Full Analysis Set | 14 |
| 8. Data for a CONSORT diagram and "study realization" | 14 |
| 9. General data | 16 |
| 9.1. Analysis set | 16 |
| 9.2. Variables | 16 |
| 9.3. Treatment of Missing and Spurious Data | 17 |
| 9.4. Exclusion of Particular Information | 17 |
| 9.5. Descriptive Analyses | 17 |
| 9.6. Hypotheses & Statistical Tests | 17 |
| 10. Primary Endpoint1 | 18 |
| 10.1. Analysis set | 18 |
| 10.2. Variables | 19 |
| 10.1. Treatment of Missing and Spurious Data | 19 |
| 10.2. Exclusion of Particular Information | 19 |
| 10.3. Descriptive Analyses | 19 |
| 10.4. Hypotheses & Statistical Tests | 19 |
| 11. Secondary Endpoint1 | 20 |
| 11.1. Analysis set | 20 |
| 11.2. Variables | 20 |
| 11.1 Treatment of Missing and Spurious Data | 21 |
| 11.2. Exclusion of Particular Information | 21 |
| 11.3. Descriptive Analyses | 21 |
| 11.4. Hypotheses & Statistical Tests | 21 |
| 12. Secondary Endpoint2 | 22 |
| 12.1. Analysis set | 22 |
| 12.2. Variables | 22 |
| 12.1. Treatment of Missing and Spurious Data | 22 |
| 12.2. Exclusion of Particular Information | 22 |
| 12.3. Descriptive Analyses | 22 |
| 12.4. Hypotheses & Statistical Tests | 22 |
| All rights pertaining to this document are exclusively held | |

BIOTRONIK excellence for life

# Statistical Analysis Plan BIO|MASTER.BIOMONITOR III Study

| _ | _ | |
|-----|-----|------|
| Paa | e : | 3/34 |

| 13. Sec | ondary Endpoint3 | 23 |
|---|---|---|
| 13.1. | Analysis set | 23 |
| 13.2. | Variables | 23 |
| 13.3. | Treatment of Missing and Spurious Data | 24 |
| 13.4. | Exclusion of Particular Information | 24 |
| 13.5. | Descriptive Analyses | 24 |
| 13.6. | Hypotheses & Statistical Tests | 24 |
| 14. Sec | ondary Endpoint4 | 26 |
| 14.1. | Analysis set | 26 |
| 14.2. | Variables | 26 |
| 14.3. | Treatment of Missing and Spurious Data | 26 |
| 14.4. | Exclusion of Particular Information | 26 |
| 14.5. | Descriptive Analyses | 27 |
| 14.6. | Hypotheses & Statistical Tests | 27 |
| 15. Dat | a of Interest | 28 |
| 15.1. | Analysis set | 29 |
| 15.2. | Variables | 29 |
| 15.2.1 | Data of interests derived from the insertion CRF only: | 29 |
| 15.2.2 | Data of interests derived from the insertion CRF and the FU CRFs: | 29 |
| 15.2.3 | Data of interests derived from the FU-CRFs: | 29 |
| 15.2.4 | Data of interests derived from the FU-CRFs and the CRF | |
| "Deac | tivation/Explantation" and FU | 29 |
| 15.2.5 | Data of interests derived from the CRFs "Deactivation/Explantation" only | 30 |
| 15.1. | Treatment of Missing and Spurious Data | 30 |
| 15.2. | Exclusion of Particular Information | 31 |
| 15.3. | Descriptive Analyses | 31 |
| 15.4. | Hypotheses & Statistical Tests | 31 |
| Reference | S | 33 |



# 1. Introduction

#### 1.1. Aim

The aim of this document is to provide detailed instructions on all descriptive and inferential statistical analyses for the Clinical Investigation Report (CIR)

Inferential analyses of the primary and secondary endpoint(s) as defined in this document are mandatory to be reported in the CIR.

#### 1.2. General information

The text contains verbatim excerpts from the CIP. Such excerpts are italicized with grey background; e.g.

#### CIP chapter 7.1 Objectives

This study is designed as a post-market clinical follow-up study to identify and evaluate residual risks associated with the use of the BIOMONITOR III system that are discovered or remain even after risk analysis, risk mitigation and successful conformity assessment. The results will be used to update the clinical evaluation. Furthermore, the study will also provide additional data as required by regulatory authorities outside of the CE-region.

The main aspects and the design of the clinical investigation are presented in chapters 0-4. General statistical procedures are summarized in chapter 5. Those methods are used in case there is no other instruction within this document.

Definitions of the specific dates, e.g. effective randomization and termination are presented in chapter 6.

Specific analysis sets are defined in chapter 0.

Descriptive and inferential statistical analyses are handled in following chapters.

Thereby the following statistical considerations are specified:

- Definition of the analysis set for the following analyses, e.g. excluding patients without any measured or imputed data for this endpoint.
- Definition of the endpoint(s) to be analyzed including references to the source data, e.g. CRF sheet and item.
- Treatment of missing and spurious data for evaluation of the above endpoint(s).
- Exclusion of particular information from the evaluation of the above endpoint(s) in addition to the exclusion of patients from the analysis set.
- Descriptive analyses including tables and figures
- Statistical alternative hypothesis/hypotheses (HA) to analyze the above endpoint(s) if available.
- Statistical tests intended to analyze the above hypothesis/hypotheses if available.



All variables are defined in tables using the following columns:

Data file
 Name of a data file exported from the CDMS with one data row per unique identifier (e.g. patient specific "patient\_display\_ID\_full") additionally, a new data file ("data\_SAR") is generated by merging all relevant data from the original CDMS data files and generating derived variables (e.g. BMI from weight and height or date of first AE episode)

Descriptive Information whether data has to be presented with descriptive methods as defined in the following sub-chapter ("Yes") or data product for generating of derived variables only ("Ne").

data needed for generating of derived variables only ("No")

• Variable name Original name of a variable in the CDMS data file or

name of a derived variables (indicated with a suffix "\_SAR");

• Variable label Original labels from the CDMS data will be used for generating the SAR

unless a new label is defined in this document ("NEW"); labels might be omitted or shortened ("...") if remaining clear

• Variable level Nominal, ordinal, scale (metric, continuous), or date

• Nominal values Original values from CDMS data will be used for generating the SAR

unless new nominal values are defined in this document ("NEW"); values might be omitted or shortened ("...") if remaining clear;

for numeric data this information is not applicable (n.a.)

| Data file, identifier | Descriptive | Variab <b>l</b> e | Variab <b>l</b> e | <b>V</b> ariab <b>l</b> e | Nominal |
|---|---|---|---|---|---|
| patient_display_id_full | | name | label | level | values |



# 2. Objectives

#### CIP chapter 7.1 Objectives

This study is designed as a post-market clinical follow-up study to identify and evaluate residual risks associated with the use of the BIOMONITOR III system that are discovered or remain even after risk analysis, risk mitigation and successful conformity assessment. The results will be used to update the clinical evaluation. Furthermore, the study will also provide additional data as required by regulatory authorities outside of the CE-region.

# 3. Investigational Device

#### CIP chapter 4 Investigational device

The devices used in this clinical investigation are the following BIOTRONIK devices:

- BIOMONITOR III incl. Incision Tool and Insertion Tool (FIT OneStep)
- Programmer devices ICS 3000 or Renamic
- Programmer Software PSW 1901.A/S
- CardioMessenger (different models)
- Remote Assistant III

# 4. Study Design & Time Course

#### CIP chapter 8.1 General considerations

The BIO\MASTER.BIOMONITOR III is designed as an open, prospective, single arm, non-randomized international study.

#### CIP chapter 8.1.4 Methods

During the course of the study, all clinical procedures are performed according to clinical routine. All parameters and measurements that are recorded within the study are described in this section and are documented on the following electronic Case Report Forms (eCRFs). The corresponding time schedule is described in section 9.1:

- Enrollment
- Baseline
- Medical History
- Insertion
- 1st follow-up
- 3-month follow-up
- 12-month follow-up
- Adverse Event
- Device Deficiency

All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.



- Device Log
- Explantation/Deactivation
- Concomitant Medication Log
- Deviation Log (site)
- Device Accountability Details (for Australia only)
- Termination



# 5. General Statistical Procedures

### 5.1. Descriptive analyses

CIP chapter ...

...

For continuous variables descriptive statistics (mean, standard deviation, minimum, 1. quartile, median, 3. quartile and maximum) will be calculated. For nominal variables absolute numbers and relative frequencies based on the non-missing data will be determined. Ordinal data are described by the 1st quartile, median, and 3rd quartile as well as the absolute numbers and relative frequencies based on the non-missing data of each category.

For illustration, see the following standard tables with and without subgroup analyses based on dummy data.

#### Nominal - dichotomous data

| Variable<br>(N total = 10) | | Category | N non-<br>missing | Absolute frequency | Relative<br>frequency<br>[%] |
|---|---|---|---|---|---|
| Sex | | Female | 9 | 5 | 55.6 |
| History of AF | | Yes | 8 | 4 | 50.0 |
| Variable<br>(N total = 10) | Category | Group<br>Randomization<br>group | N non-<br>missing | Absolute frequency | Relative<br>frequency<br>[%] |
| Sex | Female | Control<br>(N group = 3) | 3 | 2 | 66.7 |
| | | Therapy 1<br>(N group = 4) | 4 | 3 | 75.0 |
| | | All | 9 | 5 | 55.6 |
| History of AF | Yes | Control | 2 | 0 | 0.0 |
| | | Therapy 1 | 4 | 3 | 75.0 |

#### Nominal data - more than two categories

| Variable (N total = 10) Patient self assessment at enrollment Patient self assessment at 12m FU | | N non-<br>missing | Very good<br>N(%) | Good<br>N(%) | Medium<br>N(%) | Poor<br>N(%) |
|---|---|---|---|---|---|---|
| | | 7 | 2 (28.6%) | 2 (28.6%) | 1 (14.3%) | 2 (28.6%) |
| | | 8 | 1 (12.5%) | 3 (37.5%) | 3 (37.5%) | 1 (12.5%) |
| Variable<br>(N total = 10) | Group<br>Randomization<br>group | N non-<br>missing | Very good<br>N(%) | Good<br>N(%) | Medium<br>N(%) | Poor<br>N(%) |
| Patient self assessment at enrollment | Control<br>(N group = 3) | 2 | 1 (50.0%) | 0 (0.0%) | 0 (0.0%) | 1 (50.0%) |
| | Therapy 1<br>(N group = 4) | 3 | 0 (0.0%) | 1 (33.3%) | 1 (33.3%) | 1 (33.3%) |
| | All | 7 | 2 (28.6%) | 2 (28.6%) | 1 (14.3%) | 2 (28.6%) |
| Patient self assessment at 12m FU | Control | 2 | 0 (0.0%) | 1 (50.0%) | 1 (50.0%) | 0 (0.0%) |
| | Therapy 1 | 4 | 0 (0.0%) | 2 (50.0%) | 1 (25.0%) | 1 (25.0%) |
| | All | 8 | 1 (12.5%) | 3 (37.5%) | 3 (37.5%) | 1 (12.5%) |



50.0

### Scale / metric data

| Variable<br>(N total = 10) | N non-<br>missing | Mean | SD | Min | Lower quartile | Median | Upper<br>quartile | Max |
|---|---|---|---|---|---|---|---|---|
| Age [years] | 7 | 51.7 | 15.0 | 25.0 | 40.0 | 57.0 | 60.0 | 70.0 |
| Height [cm] as measured at enrollment | 8 | 177.3 | 14.4 | 150.0 | 170.0 | 179.0 | 187.5 | 195.0 |

| Variable<br>(N total = 10) | Group<br>Randomization<br>group | N non-<br>missing | Mean | SD | Min | Lower<br>quartile | Median | Upper<br>quartile | Max |
|---|---|---|---|---|---|---|---|---|---|
| Age [years] | Control<br>(N group = 3) | 2 | 55.0 | 7.1 | 50.0 | 50.0 | 55.0 | 60.0 | 60.0 |
| | Therapy 1<br>(N group = 4) | 3 | 56.7 | 15.3 | 40.0 | 40.0 | 60.0 | 70.0 | 70.0 |
| | All | 7 | 51.7 | 15.0 | 25.0 | 40.0 | 57.0 | 60.0 | 70.0 |
| Height [cm] as measured at enrollment | Control | 3 | 183.3 | 10.4 | 175.0 | 175.0 | 180.0 | 195.0 | 195.0 |
| | Therapy 1 | 3 | 175.0 | 21.8 | 150.0 | 150.0 | 185.0 | 190.0 | 190.0 |
| | All | 8 | 177.3 | 14.4 | 150.0 | 170.0 | 179.0 | 187.5 | 195.0 |

### Ordinal data

| Variable<br>(N total = 10) | N<br>missing | Min | Lower<br>quartile | Median | Upper<br>quartile | Max |
|---|---|---|---|---|---|---|
| NYHA dass enrollment | 2 | 1.0 | 1.0 | 1.0 | 2.5 | 4.0 |
| NYHA dass 24m | 3 | 1.0 | 1.0 | 1.0 | 3.0 | 4.0 |

| Variable<br>(N total = 10) | Group<br>Randomization<br>group | N non-<br>missing | Min | Lower<br>quartile | Median | Upper<br>quartile | Max |
|---|---|---|---|---|---|---|---|
| NYHA dass enrollment | Control<br>(N group = 3) | 3 | 1.0 | 1.0 | 1.0 | 3.0 | 3.0 |
| | Therapy 1<br>(N group = 4) | 4 | 1.0 | 1.0 | 1.5 | 3.0 | 4.0 |
| | All | 8 | 1.0 | 1.0 | 1.0 | 2.5 | 4.0 |
| NYHA dass 24m | Control | 2 | 1.0 | 1.0 | 2.0 | 3.0 | 3.0 |
| | Therapy 1 | 3 | 1.0 | 1.0 | 2.0 | 4.0 | 4.0 |
| | All | 7 | 1.0 | 1.0 | 1.0 | 3.0 | 4.0 |



#### 5.2. Inferential analyses

For the primary endpoint, a one-sample one-tailed binomial test will be carried out. Furthermore, a 95% confidence interval (Wilson-score method) for the SADE-free rate will be calculated. Hence, a Kaplan-Meier curve will be plotted.

Since all secondary endpoints are hypothesis-free, no inferential statistics will be carried out. Nonetheless, 95% confidence intervals for the respective parameters will be calculated.

#### 5.3. Significance level

CIP chapter 11.3: Level of significance and the power of the study

The significance level alpha is 0.025, the power is set to 90%.

A one-sided p-value < 0.025 is considered to indicate statistical significance. No adjustment for multiple testing is foreseen, i.e. all analyses except those related to the primary endpoint are considered to be exploratory.

#### 5.4. Missing Data

CIP chapter 11.11 Handling of missing, unused and spurious data

Missing or spurious data will not be imputed and not be used for analysis. More details will be specified in the SAP.

Missing data will not be imputed. Free text will be used to clarify other data. Spurious data will be clarified via the query management, i.e. corrected after approval of an investigator. Remaining outliers will be identified during the review of the data before data base closure and will be reported in the Blind Review Report. In case of a clear evidence of a measurement error, the Statistical Analysis Plan will be updated in order to avoid any bias. Spurious data, which were not clarified by the query process before database closure, will be indicated. If appropriate, analyses will be performed both with /without such data.

#### 5.5. Exclusion of data from confirmatory data analysis

CIP chapter 11.12 Exclusion of data from the confirmatory data analysis

In the following cases, data are to be excluded from analysis of the primary endpoint:

- •No data are allowed to be collected and included in the absence of a documented consent.
- •Data of patients will be excluded from analysis in case a patient terminates the study prior to any insertion attempt.



- •Patients without primary endpoint but premature study termination earlier than 77 days after insertion (91 days = 3 month minus 14 days tolerance) are not included in the analysis set to avoid an over-estimation of the SADE-free rate.
- •Any event that occurred later than the pre-specified time window for the 3-month follow-up in patients who did not have a 3-month follow-up (91 days plus 14 days tolerance = 105 days) does not contribute to the primary endpoint.
- •SADEs will be adjudicated by an internal adjudication board, whereby the investigator assessment of seriousness and device relatedness will be re-examined.

The analysis will use all data that are stored in the study database. It is in the responsibility of the persons entering data and of those checking data before the final data export that the data comply with the approval of the patient.

# 5.6. Subgroups

CIP chapter 11.9 Specification of subgroups

No subgroups are defined.

# 5.7. Interim analyses

#### CIP chapter 11.6: Provisions for an interim analysis

The main differences between BioMonitor 2 and BIOMONITOR III are limited to a reduced device size and a novel simplified injection-like insertion procedure. The focus of this study is primarily on the safety of the BIOMONITOR III system including the insertion procedure.

Therefore the primary endpoint is to evaluate the SADE-free rate related to the BIOMONITOR III and the incision and insertion tool set from insertion until the 3-month follow-up. When all enrolled patients have either completed the 3-month follow-up or their study participation has been terminated, the data for the primary endpoint are completed. At this point in time, an interim Clinical Investigation Report will be written. The content of this report will be predefined in a Statistical Analysis Plan.

Individual data collected in this study, which do not concern the primary endpoint, may be analysed before the study is completed. If they shall be published, the stipulations of section 21 apply. Safety reasons, the support of regulatory submissions and publication opportunities may trigger unscheduled interim analyses.

Such unplanned interim analyses and reports, if any, will contain at least descriptive statistics of baseline and insertion data and descriptive statistics of the defined endpoints. Inferential statistics of endpoints may be included to support publication activities. The precise scope of each interim analysis will be defined in the SAP before the individual interim analyses.

In case of a suspension of the clinical investigation, an interim analysis will be performed to generate a clinical investigation report according to the MDR requirements. No multiplicity adjustment is foreseen.



# 5.8. Software

All analyses will be carried out using validated software, e.g. SAS version 9.4 or upgrades.



# **6. Specific Study Dates**

#### 6.1. Enrollment date

| Data file, identifier | Variab <b>l</b> e | Variab <b>l</b> e | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| enrollment | DMICDT | Patient: Date of IC signature | date | n.a. |

#### 6.2. Insertion date

| Data file, identifier | Variable | Variab <b>l</b> e | Variable | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| insertion | PRIMSTDT | Date of insertion procedure | date | n.a. |

#### 6.3. Termination date

| Data file, identifier | Variab <b>l</b> e | Variable | Variab <b>l</b> e | Nominal |
|---|---|---|---|---|
| patient_display_id_full | name | label | level | values |
| termination | DSTRDT | Date of study termination | date | n.a. |



# 7. Analysis Sets

# 7.1. Full Analysis Set



| Data file,<br>identifier patient_<br>display_id_full | Variable<br>name | Variable<br>label | Variable<br>Level | Nominal<br>values | Notes |
|---|---|---|---|---|---|
| enrollment | DMSUBSPS | Patient signed the informed consent personally | Nominal | Yes<br>No | |
| enrollment | DMRPRSPS | An independent witness signed the informed consent since the patient is unable to write | Nominal | Yes<br>No | |
| dataSAR | full_set_sar | All patients | Nominal | Yes<br>No | |



# 8. Data for a CONSORT diagram and "study realization"

The following data shall be reported:

- Number of patients with enrollment data
- Number of enrollments per site
- Date of FPI, LPI, LPO per site and total
- Cumulative and mean/median FU duration from insertion to last available CRF information
- Cumulative and mean/median FU duration from enrollment to termination date on termination CRF

The following variables will be calculated:

| Data file, identifier patient_ display_id_full | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|
| | name | label | Level | values |
| insertion | PRIMSTDT | Date of insertion | date | n.a. |





| enrollment | dmicdt | Date of informed consent | date | n.a. |
|---|---|---|---|---|
| Follow-up_1st | svstdt -><br>svstdt_fu1 | Date of visit 1. FU | date | n.a. |
| Follow-up_3months | svstdt -><br>svstdt_fu3m | Date of visit 3 months FU | date | n.a. |
| Follow-up_12months | svstdt -><br>svstdt_fu12m | Date of visit 12 months FU | date | n.a. |
| hospitalization_log | hostdt | Hospitalization Start date | date | n.a. |
| data_sar | sar_hospstdt_first1 | onset date of first hosp. | date | n.a. |
| data_sar | sar_hospendt_last <sup>2</sup> | date of resolution/death of last AE | date | n.a. |
| adverse_event | aestdt | Onset Date of AE | date | n.a. |
| data_sar | sar_aestdt_first <sup>3</sup> | onset date of first AE | date | n.a. |
| data_sar | sar_aeendt_last <sup>4</sup> | date of resolution/death of last AE | date | n.a. |
| termination | dstrdt | Date of study termination | date | n.a. |
| data_SAR | sar_last_crf <sup>5</sup> | Date of last CRF information | date | n.a. |
| data_SAR | sar_time_crf <sup>6</sup> | time [days] from insertion to last CRF | scale | |
| data_SAR | sar_time_term <sup>7</sup> | time [days] from insertion to termination | scale | |
| data_SAR | sar_time_max <sup>8</sup> | time [days] from insertion to termination or last CRF | scale | |

For all patients with premature study duration or missing insertion or any violation of in-/exclusion criteria the following variables shall be listed:

- All in-/exclusion criteria
- Date of enrollment
- Date and reason of premature study termination
- Date and type of all other available CRFs (except for AE-CRFs)





# 9. General data

# 9.1. Analysis set

All analyses are performed for the full analysis set<sup>9</sup>.

### 9.2. Variables



### 9.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4

#### 9.4. Exclusion of Particular Information

See general definitions in chapter 5.5

No data are excluded from the analysis from the above analysis set and variables.

### 9.5. Descriptive Analyses

See general definitions in chapter 5.1 and exceptions for reporting numbers and text below the variable tables, if appropriate.

### 9.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



# 10. Primary Endpoint1

CIP chapter 7.2.1 - Primary endpoint and hypothesis

SADE-free rate until the 3-month follow-up

A primary endpoint is an SADE (see definition in section 18) that is possibly, probably or causally related to the BIOMONITOR III, the Incision Tool or the Insertion Tool, or the insertion procedure, which occurs before the 3-month follow-up.

SADEs will be adjudicated by an internal adjudication board, whereby the seriousness and device relatedness will be re-examined. If any amply documented external physical influence (e.g. accident, sport) or medical AE caused the SADE, it does not contribute to this endpoint. SADEs that occur later than the 3-month follow-up, and SADEs with onset date later than 105 days after insertion procedure (3 months defined as 91 days after implantation + 14 days would still be in accordance to the CIP) in case the 3-month follow-up was not conducted or conducted outside the specified time interval, do not contribute to this endpoint.

The parameter of interest is the SADE free rate, which will be calculated by

Number of patients with one or more primary endpoint until the 3 months FU

Number of patients at the 3 months FU or with primary endpoint

in percent. The period of observation starts with the insertion of the BIOMONITOR III and takes until the 3-month follow-up.

#### 10.1. Analysis set

The number of patients with at least one primary endpoint until the 3 months FU (the numerator) will be determined by assessing the variable "AERELPET" in the "AE evaluation" form. This form is filled by the AE evaluation board and the variable "AERELPET" is set to "Yes" if and only if all conditions defined in 7.2.1 in the CIP are met.

The denominator will be calculated as follows:

- 1. The number of patients with 3 months FU will be counted by the number of non-missing entries in SVSTDT in the "3 month FU" form.
- 2. The number of patients with primary endpoint will be calculated as defined above.
- 3. In case of patients lying in the intersection of both sets, these patients will be counted once.
- 4. Patients without SADE and termination date less than 77 days after insertion will be disregarded.

Patients who do not attend the 3 months FU, but who have not terminated study participation earlier than 77 days after insertion will be included in the analysis.

For the calculation of the Kaplan-Meier analysis, the following time variables will be used:

- 1. For patients with at least one primary endpoint: time from insertion to time of first primary endpoint
- 2. For patients without primary endpoint: time from insertion to last information available

BIOTRONIK excellence for life

For the KM analysis data of all patients is used.

#### 10.2. Variables

| Data file,<br>identifier patient_<br>display_id_full | Notes | | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|---|
| AE evaluation | sorted by<br>patient_<br>display_id_<br>full and<br>AESTDT<br>and<br>removed<br>duplicates | | Adverse event is relevant for primary endpoint | nominal | Yes<br>No |
| 3-month FU | | SVSTDT | Date of visit | date | |
| 3-month FU | | sar_3mFU_available | 3m FU available? | nominal | Yes<br>No |
| Termination | | | Termination less than 77 days after insertion? | nominal | Yes<br>No |

#### 10.1. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4

#### 10.2. Exclusion of Particular Information

See general definitions in chapter 5.5

No data are excluded from the analysis from the above analysis set and variables.

# 10.3. Descriptive Analyses

See general definitions in chapter 5.1 and exceptions for reporting numbers and text below the variable tables, if appropriate.

Furthermore a Kaplan-Meier analysis (including Kaplan-Meier plot) will be calculated and the estimation of the SADE-free rate (including two-sided 95% confidence interval) at 3 months (= 90 days) will be given.

# 10.4. Hypotheses & Statistical Tests

Null hypothesis:  $H_{0}: p_{SADE} \leq 90\%$ 

Alternative hypothesis:  $H_A: p_{SADE} > 90\%$ 

The hypothesis will be tested by using an exact binomial test against the value of 0.9. An exact two-sided confidence interval for the SADE-free rate.



# 11. Secondary Endpoint1

#### CIP chapter 7.2.2: Secondary endpoints

#### R-wave amplitude

The secondary endpoint 1 evaluates the R-wave amplitude at the 1st follow-up and at 3-month follow-up by measuring both, the lowest and the highest amplitude value via the programmer.

The secondary endpoint "R-wave amplitude" will be calculated as the mean value from the lowest and the highest amplitude.

### 11.1. Analysis set

All analyses are performed for the full analysis set12.

#### 11.2. Variables

| Data file,<br>identifier patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level |
|---|---|---|---|---|
| insertion | | DUHLRWA -><br>DUHLRWA ins | Highest amplitude<br>value [mV] | Scale |
| insertion | | DULLRWA -><br>DULLRWA_ins | lowest amplitude<br>value [mV] | Scale |
| insertion | | DULRWA_ins_m <sup>13</sup> | mean of highest and lowest value [mV] | Scale |
| follow_up_1st | | DUHLRWA -><br>DUHLRWA_fu1 | Highest amplitude value [mV] | Scale |
| follow_up_1st | | DULLRWA -><br>DULLRWA_fu1 | lowest amplitude value [mV] | Scale |
| follow_up_1st | | DULRWA_fu1_m <sup>14</sup> | mean of highest and lowest value [mV] | Scale |
| follow_up_3months | | DUHLRWA -><br>DUHLRWA_fu3 | Highest amplitude value [mV] | Scale |
| follow_up_3months | | DUHLRWA -><br>DULLRWA_fu3 | lowest amplitude value [mV] | Scale |
| follow_up_3months | | DULRWA_fu3_m <sup>15</sup> | mean of highest and lowest value [mV] | Scale |
| follow_up_12months | | DUHLRWA -><br>DUHLRWA_fu12 | Highest amplitude value [mV] | Scale |
| follow_up_12months | | DUHLRWA -><br>DULLRWA_fu12 | lowest amplitude value [mV] | Scale |
| follow_up_12months | | DULRWA_fu12_m <sup>16</sup> | mean of highest and lowest value [mV] | Scale |







# 11.1. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4

#### 11.2. Exclusion of Particular Information

No data are excluded from the analysis from the above analysis set and variables.

# 11.3. Descriptive Analyses

See general definitions in chapter 5.1 and exceptions for reporting numbers and text below the variable tables, if appropriate.

In addition, boxplots will be generated.

### 11.4. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



# 12. Secondary Endpoint2

CIP chapter 7.2.2: Secondary endpoints

#### Noise burden

The secondary endpoint 2 evaluates the noise burden at the 1st follow-up and at 3-month follow-up by retrieving the percentage of noise via the programmer.

#### 12.1. Analysis set

All analyses are performed for the full analysis set<sup>17</sup>.

#### 12.2. Variables

| Data file,<br>identifier patient_<br>display_id_full | Notes | | | 1 | Nominal<br>values |
|---|---|---|---|---|---|
| follow_up_1st | | DUNSE | Noise [%] | Scale | |
| follow_up_3months | | DUNSE | Noise [%] | Scale | |
| follow_up_12months | | DUNSE | Noise [%] | Scale | |

Moreover, the proportions of patients with "Noise smaller 5% vs. at least 5%" will be reported for the 1 month FU, 3 months FU and 12 months FU separately and in total (all FU together). Therefore the variable "DUNSE" will be recoded accordingly.

#### 12.1. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4

#### 12.2. Exclusion of Particular Information

No data are excluded from the analysis from the above analysis set and variables.

#### 12.3. Descriptive Analyses

See general definitions in chapter 5.1 and exceptions for reporting numbers and text below the variable tables, if appropriate.

In addition, boxplots will be generated.

### 12.4. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



# 13. Secondary Endpoint3

CIP chapter 7.2.2: Secondary endpoints

Assessment of P-wave visibility

The secondary endpoint 3 evaluates the P-wave visibility at 1st, 3- and 12-month follow-up. The investigator will evaluate whether P-waves can be recognized in the stored sECGs showing sinus rhythm. The number of heart cycles and observed P-waves which can undoubtly be identified in ECGs will be assessed by the investigator.

### 13.1. Analysis set

All analyses are performed for the full analysis set18.



### 13.2. Variables

| Data file,<br>identifier patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| follow_up_1st | | EGCCCNUM01 | Exact number of cardiac cycles | Scale | |
| follow_up_1st | | EGPWNUM01 | Exact number of clearly identifiable P-waves | Scale | |
| sar_data | | sar_pwavevis_fu1_1 | P-wave visibility FU1 1st [%] | | |
| follow_up_1st | | EGCCCNUM02 | Exact number of cardiac cycles | Scale | |
| follow_up_1st | | EGPWNUM02 | Exact number of clearly identifiable P-waves | Scale | |
| sar_data | | sar_pwavevis_fu1_2 | P-wave visibility FU1 2nd [%] | | |
| sar_data | | sar_pwavevis_fu1_t<br>ot <sup>21</sup> | P-wave visibility pooled [%] | | |





| follow_up_3months | EGCCCNUM -> | Exact number of cardiac | Scale |
|---|---|---|---|
| | EGCCCNUM_3m | cycles | |
| follow_up_3months | EGPWNUM -> | Exact number of clearly | Scale |
| | EGPWNUM_3m | identifiable P-waves | |
| sar_data | sar_pwavevis_fu3 <sup>22</sup> | P-wave visibility 3m [%] | |
| follow_up_12month | EGCCCNUM -> | Exact number of cardiac | Scale |
| S | EGCCCNUM_12m | cycles | |
| follow_up_12month | EGPWNUM -> | Exact number of clearly | Scale |
| s | EGPWNUM_12m | identifiable P-waves | |
| car data | sar_pwavevis_fu12 | P-wave visibility 12m | |
| sar_data | 23 | [%] | |
| car data | sar_pwavevis_tot <sup>24</sup> | P-wave visibility total | |
| sar_data | | [%] | |

# 13.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4



#### 13.4. Exclusion of Particular Information

No data are excluded from the analysis of the above analysis set and variables.

Also data from the 3 months and 12 months FU which are outside the defined time range will be considered her.

#### 13.5. Descriptive Analyses

See general definitions in chapter 5.1 and exceptions for reporting numbers and text below the variable tables, if appropriate.

In addition, boxplots will be generated.

Moreover, the rate of patients with a P-wave visibility of at least 5% shall be reported for each follow-up separately and the number of patients with a P-wave visibility of at least 5% at all available follow-ups shall be reported.

#### 13.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.





# 14. Secondary Endpoint4

CIP chapter 7.2.2: Secondary endpoints

SADE-free rate until the 12-month follow-up

The secondary endpoint 4 is the SADE-free rate related to the BIOMONITOR III 12 months after insertion.



# 14.1. Analysis set

All analyses are performed for the full analysis set<sup>25</sup>.

For the calculation of the Kaplan-Meier analysis, the following time variables will be used:

- 1. For patients with at least one primary endpoint: time from insertion to time of first primary endpoint (sar\_aestdt\_first).
- 2. For patients without primary endpoint: time from insertion to last information available (sar\_time\_max).

For the KM analysis data of all patients is used.

#### 14.2. Variables

| Data file,<br>identifier patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|---|
| AE evaluation | sorted by patient_display_id_full and AESTDT and removed duplicates | AERELPET | Adverse event is relevant for primary endpoint | nominal | Yes<br>No |

#### 14.3. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4

#### 14.4. Exclusion of Particular Information

No data are excluded from the analysis from the above analysis set and variables.



### 14.5. Descriptive Analyses

A Kaplan-Meier analysis (including Kaplan-Meier plot) will be calculated and the estimation oft he SADE-free rate (including two-sided 95% confidence interval) at 12 months (= 365 days) will be given.

# 14.6. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.



#### 15. Data of Interest

#### CIP chapter .7.5 Further data of interest

Beyond the objectives defined in section 7.1, the study is designed to collect further data of interest. The data on the following topics will be considered `data of interest´ and may be analyzed, as appropriate:

- Demographics
- Medical history
- Indication for ICM
- Usage of incision tool and assessment of incision tool handling
- Assessment of insertion procedure: performance of insertion tool and ease of use (e.g. insertion time, handling and positioning)
- Insertion site
- Insertion success rate
- Wound closure
- Positioning of BIOMONITOR III
- · Comfort after wound healing
- Explantation data of BIOMONITOR III
- Additional implantation of BIOMONITOR III
- Serial number of used study devices
- Performance of arrhythmia detection (will be assessed by comparing the BIOMONITOR III detected arrhythmia episodes recorded against a 48-hour Holter ECG, if applicable)
- Syncope and AF: detailed analysis of sensing performance in device-triggered ECGepisodes
- AF burden
- Assessment of device programming: individualized programming and re-programming of the device
- Assessment of programmer and programmer software performance
- Remote Assistant III trigger success rate after insertion procedure
- Home Monitoring Data (e.g. transmission success)
- HM workflow efficiency

Assessment of BIOMONITOR III repositioning (if applicable)

- Assessment of BIOMONITOR III migration (if applicable)
- Usability of Patient App (if applicable)
- Information on application of imaging techniques, if applicable (e.g. MRI, mammography)
- Diagnosis and further treatment
- Adverse events and device deficiencies

The topics "demographics", "medical history", and "indication for ICM" are already included in chapter 9.

"Adverse events and device deficiencies" will be reported as provided by the safety report from the vigilance department.



The topics "arrhythmia detection performance", "sensing performance in device triggered ECG episodes" and all analyses based on Home Monitoring data are beyond the scope of this document.

#### 15.1. Analysis set

All analyses are performed for the full analysis set<sup>26</sup>.

#### 15.2. Variables

#### 15.2.1 Data of interests derived from the insertion CRF only:

This includes the following data of interest:

- Usage of incision tool and assessment of incision tool handling
- Assessment of insertion procedure: performance of insertion tool and ease of use (e.g. insertion time, handling and positioning)
- · Insertion site
- Insertion success rate
- Wound closure
- Positioning of BIOMONITOR III
- Remote Assistant III trigger success rate after insertion procedure (for all patients and split by BMI with a cut-off of 30)
- Assessment of BIOMONITOR III repositioning (if applicable)



#### 15.2.2 Data of interests derived from the insertion CRF and the FU CRFs:

This includes the following data of interest:

- Assessment of device programming: individualized programming and re-programming of the device
- Assessment of programmer and programmer software performance

#### 15.2.3 Data of interests derived from the FU-CRFs:

This includes the following data of interest:

- Comfort after wound healing
- Usability of Patient App (if applicable)
- Information on application of imaging techniques, if applicable (e.g. MRI, mammography)

# 15.2.4 Data of interests derived from the FU-CRFs and the CRF "Deactivation/Explantation" and FU

This includes the following data of interest:

Assessment of BIOMONITOR III migration (if applicable)I



#### 15.2.5 Data of interests derived from the CRFs "Deactivation/Explantation" only

This includes the following data of interest:

- Explantation data of BIOMONITOR III
- Diagnosis and further treatment
- Additional implantation of BIOMONITOR III

In addition to the descriptive reporting of the parameters related to diagnosis and further treatment, a case-by-case listing shall be provided for all patients with a deactivation or explantation. This listing shall contain the following variables:

#### Baseline CRF:

| CEINDICM | Primary type of ICM indication |
|----------|-------------------------------------------------------|
| COINDICM | Specification of other primary type of ICM indication |

#### Deactivation/Explantation CRF:

| DXEXREA | Reason for explantation/deactivation |
|----------|---------------------------------------------------------|
| PRDGNDT | Date of diagnosis |
| DUBMDGN | Did the BIOMONITOR III contribute to this diagnosis? |
| DUBMDGNA | How did the BIOMONITOR III contribute to the diagnosis? |
| CVARTYP | Specify arrythmia type detected |
| QSFTRT01 | Ablation procedure |
| QSABPR | Specify the ablation procedure |
| QSFTRT02 | Medication |
| QSCM01 | Anticoagulation |
| QSCM02 | Antiarrhythmics |
| QSCMOTH | Other |
| QSFTRT03 | ICD implantation |
| QSFTRT04 | Pacemaker implantation |
| QSFTRTOT | Other |
| QSBMU | Further use of the BIOMONITOR III |

#### 15.1. Treatment of Missing and Spurious Data

See general definitions in chapter 5.4



#### 15.2. Exclusion of Particular Information

See general definitions in chapter 5.5

No data are excluded from the analysis from the above analysis set and variables.

#### 15.3. Descriptive Analyses

See general definitions in chapter 5.1 and exceptions for reporting numbers and text below the variable tables, if appropriate.

### 15.4. Hypotheses & Statistical Tests

There are no pre-defined statistical hypotheses.







# References

References for specific statistical procedures



### **Abbreviations**

ADE Adverse Device Effect

AE Adverse Event
AF Atrial Fibrillation

CDMS Clinical Data Management System

CI Confidence Interval

CIP Clinical Investigation Plan
CIR Clinical Investigation Report

CRF Case Report Form

FU Follow-up

SADE Serious Adverse Device Event

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAR Statistical Analysis Report
SOP Standard Operating Procedure

SD Standard Deviation

